CLINICAL TRIAL: NCT06782945
Title: A Direct-to-Consumer Placebo-controlled Study Investigating the Effectiveness of 2 Different Doses of BIOHM FX Probiotic Blend in Improving Digestive Symptoms in Individuals With Moderate Gastrointestinal Discomfort
Brief Title: Investigating the Effectiveness of 2 Different Doses of BIOHM FX Probiotic Blend in Improving Digestive Symptoms
Status: Active, not recruiting | Type: Observational
Sponsor: Biohm Technologies (Industry)
Collaborators: People Science, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PS09
Record Dates: First submitted 2024-11-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Moderate Gastrointestinal Discomfort

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BIOHM FX Probiotic Blend 1 billion CFU: Participants will be randomized to one of 3 groups: (1) BIOHM FX Probiotic Blend 1 billion CFU, (2) BIOHM FX Probiotic Blend 3 billion CFU, and (3) Matching placebo. The Investigators and study team and Participants will be blinded to the group assignment. Screening assessments, questionnaires, scales, surveys, and at-home stool collection during the use of the study product/placebo and end of study experience survey data will be collected.
  Interventions: Dietary Supplement: BIOHM FX Probiotic Blend
- BIOHM FX Probiotic Blend 3 billion CFU: Participants will be randomized to one of 3 groups: (1) BIOHM FX Probiotic Blend 1 billion CFU, (2) BIOHM FX Probiotic Blend 3 billion CFU, and (3) Matching placebo. The Investigators and study team and Participants will be blinded to the group assignment. Screening assessments, questionnaires, scales, surveys, and at-home stool collection during the use of the study product/placebo and end of study experience survey data will be collected.
  Interventions: Dietary Supplement: BIOHM FX Probiotic Blend
- Placebo: Participants will be randomized to one of 3 groups: (1) BIOHM FX Probiotic Blend 1 billion CFU, (2) BIOHM FX Probiotic Blend 3 billion CFU, and (3) Matching placebo. The Investigators and study team and Participants will be blinded to the group assignment. Screening assessments, questionnaires, scales, surveys, and at-home stool collection during the use of the study product/placebo and end of study experience survey data will be collected.
  Interventions: Dietary Supplement: BIOHM FX Probiotic Blend

INTERVENTIONS:
Dietary Supplement: BIOHM FX Probiotic Blend — BIOHM Health has been selling BIOHM FX, a blend of probiotics as a dietary supplement addressed at the digestive health market since 2017. The blend is present in the market in various concentrations ranging from 30 Billion CFU to 1 Billion CFU. The probiotic blend consists of Lactobacillus acidophilus, Lactobacillus rhamnosus, Saccharomyces boulardii, Bifidobacterium breve and amylase. The blend is manufactured at cGMP facilities located in the United States and has attained self GRAS status. Prior to release, each lot of probiotic blend is tested for heavy metals, objectionable organisms, water content, probiotic potency, enzyme activity level and allergens, Soy, Milk and Gluten. Additionally, BIOHM performs annual testing for a full FALCPA panel of allergens ensuring there are no allergens present in the blend.

SUMMARY:
The rationale for this study is to observe the effect of two different doses of a consumer-grade probiotic product called FX Probiotic Blend on digestive symptoms in individuals with moderate gastrointestinal discomfort. Additionally, the study aims to observe the effects of the probiotic product on anxiety and quality of life, as well as effects on gut microbiota via activities and technologies that can successfully and effectively be completed and utilized in a home setting. Because this product is currently available in the overt the counter (OTC) market across the United States, a consumer-driven, decentralized observational clinical research study is therefore well-suited for examining the effects of this probiotic product in this population.

DETAILED DESCRIPTION:
Digestive health has garnered significant attention among consumers as evidenced by the 2012 National Health Initiative Survey (NHIS) reporting approximately 4 million adults using dietary supplements aimed at enhancing digestive wellness. Probiotics which are beneficial bacteria and yeast primarily residing in the gastrointestinal tract are available as dietary supplements and are present in naturally occurring foods such as yogurt, kefir, sauerkraut, tempeh and kimchi. Previous research indicates improved digestive health, immune boosting and improved mental health, yet further investigation is warranted. This study aims to assess the impact of oral supplementation with a probiotic blend on gastrointestinal symptoms and alterations in microbiome composition.

BIOHM Health has been selling BIOHM FX, a blend of probiotics as a dietary supplement addressed at the digestive health market since 2017. The blend is present in the market in various concentrations ranging from 30 Billion colony forming units (CFU) to 1 Billion colony forming units (CFU). The probiotic blend consists of Lactobacillus acidophilus, Lactobacillus rhamnosus, Saccharomyces boulardii, Bifidobacterium breve and amylase. The blend is manufactured at Current Good Manufacturing Practice (cGMP) facilities located in the United States and has attained self Generally Recognized as Safe (GRAS) status. Prior to release, each lot of probiotic blend is tested for heavy metals, objectionable organisms, water content, probiotic potency, enzyme activity level and allergens, Soy, Milk and Gluten. Additionally, BIOHM performs annual testing for a full Food Allergen Labeling and Consumer Protection Act (FALCPA) panel of allergens ensuring there are no allergens present in the blend.

BIOHM FX has previously been studied to show a number of digestive health-related properties such as supporting healthy digestion, reduced bloating, flatulence, abdominal pain and constipation. Additionally BIOHM FX has been shown to break down polymicrobial biofilms, and support healthy candida levels.

The rationale for this study is to observe the effect of two different doses of a consumer-grade probiotic product called FX Probiotic Blend on digestive symptoms in individuals with moderate gastrointestinal discomfort. Additionally, the study aims to observe the effects of the probiotic product on anxiety and quality of life, as well as effects on gut microbiota via activities and technologies that can successfully and effectively be completed and utilized in a home setting. Because this product is currently available in the over the counter (OTC) market across the United States, a consumer-driven, decentralized observational clinical research study is therefore well-suited for examining the effects of this probiotic product in this population.

The study team will examine the outcomes in a broad age-range of adults who have chosen to try this product. The study will incorporate participant reported outcome questionnaires and surveys and at-home stool collection. There is no "doctor-patient" relationship as part of this research since the participant as a consumer is making the informed choice to take the product and take part in the observational process with self-reported measures and at-home sample collection. Findings from this study will contribute knowledge toward the dosing and formulation of the probiotic product and the design of future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75 years old, inclusive
* Has self-reported moderate digestive symptoms, such as abdominal pain, bloating, flatulence, constipation, or diarrhea.
* Has a moderate Gastrointestinal Symptom Rating Scale (GSRS) score between 4-5.
* Willingness to refrain from taking probiotics or prebiotics during the study period.
* Interested in understanding more about their gut health and the use probiotic products
* If taking any OTC or prescription medications for anxiety (e.g. magnesium, anticholinergics, Buspirone, Tricyclics, MAOIs,) or other class of medication for anxiety, must be on a stable dose for at least 4 weeks prior to randomization and throughout the course of the study.
* If using any cannabis-containing products, must be on a stable regimen for at least 4 weeks prior to randomization and throughout the course of the study.
* If using any nicotine-containing products, must be on a stable regimen for at least 4 weeks prior to randomization and throughout the course of the study.
* In good general health at the time of screening (Investigator discretion).
* Able to read and understand English.
* Able to read, understand, and provide informed consent.
* Able to use a personal smartphone device and download Chloe by People Science.
* Able to receive shipment of the product at an address within the United States.
* Able to complete study assessments over the course of up to 7 weeks.

Exclusion Criteria:

* Do not have a personal smartphone, internet access, or unwilling to download Chloe.
* Concomitant Therapies:

  * Participants receiving any investigational therapies or treatments within 30 days prior to randomization.
  * Participants currently taking or have taken antibiotics, probiotics, or prebiotics within the past 4 weeks prior to randomization.
  * Participants using immunosuppressive medications, systemic steroids, antifungals or other medications known to significantly impact gastrointestinal function or microbiota.
* Other Illnesses or Conditions: Participants who have the following comorbidities or gastrointestinal illnesses are excluded:

  --Participants with a clinical diagnosis of any gastrointestinal illness, including but not limited to:
* Inflammatory bowel disease (Crohn's disease, ulcerative colitis)
* Gastroesophageal reflux disease (GERD)
* Gastric or duodenal ulcers
* Celiac disease
* Diverticular disease
* Chronic pancreatitis
* Gastroparesis
* Severe liver disease (e.g., cirrhosis, hepatitis, NAFLD acceptable)
* Gallbladder disease (e.g., cholecystitis, cholelithiasis)
* Gastrointestinal cancer (Colorectal, Intestinal, Stomach, Liver, Gallbladder)
* Participants with a known or suspected gastrointestinal infection, such as:
* Clostridium difficile infection
* Helicobacter pylori infection
* Parasitic infections (e.g., Giardia, Cryptosporidium)
* Participants with a history of gastrointestinal surgery, excluding appendectomy and cholecystectomy.
* Participants with a history of gastrointestinal bleeding or perforation.
* Currently diagnosed with Alcohol Abuse and/or Substance Use Disorder
* Currently pregnant, planning to become pregnant in the next 1 month, or breastfeeding
* Willing to practice a reliable method of contraception for the duration of the study
* Any underlying medical conditions or comorbidities that may confound the assessment of digestive symptoms or the evaluation of the study outcomes.
* Have a significant illness, disease or condition which, in the opinion of the principal investigator, may impact their ability to participate in the study or impact the study outcomes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Individuals with Moderate Gastrointestinal Discomfort
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-03-04 (Estimated)

PRIMARY OUTCOMES:
To observe the effect of two different doses of BIOHM FX Probiotic blend on digestive symptoms | 6 weeks
  Change in the Gastrointestinal Symptom Rating Scale (GSRS) score between placebo and study product groups. Baseline period will be compared as well as GSRS scores between the two doses.
  The score is calculated by using a 7-point Likert scale to rate the frequency and intensity of symptoms experienced over the previous week. A higher score indicates more severe symptoms and worse outcomes.

SECONDARY OUTCOMES:
To assess the effect of two different doses of BIOHM FX Probiotic blend on gut microbiome markers | 6 weeks
  Change in gut microbiome, specifically in probiotic species of bacteria and fungi between placebo and study product groups at Week 6 as analyzed and measured from stool specimens. Baseline period will be compared as well as changes between the two doses.
  There are no minimum and maximum values as stool samples will be analyzed.
To assess the effect of two different doses of BIOHM FX Probiotic blend on anxiety | 6 weeks
  Change in Anxiety Symptom Questionnaire (ASQ) score at Week 6 between placebo and study product groups. Baseline period will be compared as well as scores between the two doses.
  Each item on the Anxiety Symptom Questionnaire is rated on a 10-point scale, assessing both the intensity and frequency of anxiety symptoms. Higher scores on the Anxiety Symptom Questionnaire indicate greater anxiety severity.
To assess the effect of two different doses of BIOHM FX Probiotic blend on gastrointestinal symptoms (i.e. flatulence, bloating, abdominal discomfort, stool consistency/ regularity, constipation) | 6 weeks
  Change in gut microbiome, specifically in opportunistic pathogenic species of bacteria and fungi at Week 6 between placebo and study product groups as analyzed and measured from stool specimens. Baseline period will be compared as well as changes between the two doses.
  There are no minimum and maximum values as stool samples will be analyzed.
To assess the effect of two different doses of BIOHM FX Probiotic blend on quality of life | 6 weeks
  Change in average scores of gastrointestinal symptoms (i.e flatulence, bloating, abdominal discomfort, stool consistency/ regularity, constipation) between placebo and study product groups as measured by daily survey questions. Baseline period will be compared as well as scores between the two doses. Change in the Short Form (SF-36) Survey, a health-related quality of life, score at Week 6 between placebo and study product groups. Baseline period will be compared as well as scores between the two doses.
  The Short Form (SF-36) Survey score is a number between 0 and 100, with higher scores indicating better health. A score of 0 indicates maximum disability, while a score of 100 indicates no disability.
To observe the safety and tolerability of two different doses of BIOHM FX Probiotic blend | 6 weeks
  Assessment of the number, frequency, and severity of adverse events (AEs), serious adverse events (SAEs) and adverse event withdrawals reported over the study product/placebo use period.
  There are no minimum and maximum values for adverse events, the more and/or serious the adverse event the worse the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Craft, MD, Principal Investigator — People Science, Inc.
Locations (1):
- People Science, Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided